CLINICAL TRIAL: NCT01231425
Title: Prospective Epidemiological Study To Evaluate The Clinical Utility Of Acupuncture In The Treatment Of Back Pain (Study PUCTURE-CV)
Brief Title: Prospective Study of Clinical Utility of Acupuncture in Back Pain
Acronym: PUCTURE-CV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Group G-6 (Network)
Responsible Party: Sponsor
Other Study IDs: GE6-ACU-2010-01
Record Dates: First submitted 2010-09-28; First posted 2010-11-01 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Back Pain; Musculoskeletal Disease
Keywords: Back pain; cervicalgia; dorsalgia; lumbalgia; acupuncture
MeSH Terms: conditions — Back Pain; Musculoskeletal Diseases; Neck Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With usual concomitant treatment: Two observational cohorts of patients will be evaluated: with and without concomitant analgesic/ antiinflammatory drugs. The objective is evaluate that both therapies (drugs and acupuncture) could be used as adjunctive therapy in order to maximize the analgesia that could be reached
- Without usual concomitant treatment: This group include patients that are not been treated with analgesic drugs at the beginning of the study. As an observational and naturalistic study any indicated treatment is allowed in any time

SUMMARY:
The purpose of this study is to evaluate prospectively the effectiveness of acupuncture as adjunctive therapy in the treatment of spinal pain is the three backbone areas: cervical, thoracic and lumbar pain, under conditions of usual clinical practice as the medical acupuncturist performed acupuncture, with and without supplementary pharmacological treatment during the first 4 weeks of follow up.

DETAILED DESCRIPTION:
Epidemiological, observational, prospective, with two cohorts, naturalistic and non-interventionist study.

The disease to be studied is Back pain (cervical, thoracic or lumbar) caused by musculoskeletal pathologies and previously treated with conventional medical treatment with or without treatment currently.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18 and over
* Patients diagnosed with back pain: cervical, thoracic or lumbar.
* Patients who has received appropriate medical treatment for their disease: analgesics, anti-inflammatories, or other treatments, but painful and symptoms persist
* Patients that could receive acupuncture treatment in order to reduce the symptoms and reviewed by a medical acupuncturist
* Patients with sufficient cultural and educational level to complete the health questionnaires required in the study
* Patients who have given their written informed consent to participate in the study

Exclusion Criteria:

* Patient with any illness and that medical opinions recommended not to participate in the study
* Patient can not respond to questionnaires administered during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients who go to the Acupuncture Office diagnosed of cervical, thoracic or lumbar pain caused by musculoskeletal diseases, pretreated with pharmacological treatment, they start treatment with acupuncture as adjunctive therapy for symptoms of their disease.
  Initially it was estimated that the optimal number of patients included to achieve the objectives of the study is 102 patients
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
VAS: Visual Analogic Scale of pain | 10 weekly visits
  Pain assesment will be evaluated using a Visual Analogic Scale of pain (VAS). This variable will be evaluated in all 10 visits and it will be showed its evolution (decrease) along the study

SECONDARY OUTCOMES:
Sheehan Disability Questionnaire | First Visit (week 1) and Final Visit (week 10)
  Sheehan Disability Questionnaire, this validated questionnaire will be administrated in Visit 1 (Basal) and Visit 10 (Final) and it will be compared if there has been statistical differences between both evaluations
Evaluation of the Scale Hospital Anxiety Depression (HAD) | First Visit (week 1) and Final Visit (week 10)
  Scale Hospital Anxiety Depression (HAD), this scale will be evaluated using a validated questionnaire administrated in Visit 1 (basal) and Visit 10 (Final) and it will be compared if there has been statistical differences between both evaluations
Health Questionnaire EuroQol-5D | First Visit (week 1) and Final Visit (week 10)
  Health Questionnaire EuroQol-5D, this validated questionnaire will be administrated in Visit 1 (Basal) and Visit 10 (Final) and it will be compared if there has been statistical differences between both evaluations
Assessment of sleep with the integrated scale MOS (Medical Outcomes Study) | First Visit (week 1) and Final Visit (week 10)
  Assessment of sleep with the integrated scale MOS (Medical Outcomes Study), this scale will be evaluated using a validated questionnaire administrated in Visit 1 (basal) and Visit 10 (Final) and it will be compared if there has been statistical differences between both evaluations
McGill Pain Questionnaire | 10 weekly visits
  A secondary evaluation of pain suffered by the patients will be evaluated using the validated McGill Pain Questionnaire. This questionnaire will be adminstrated in all 10 visits and it will be showed its evolution (decrease) along the study

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Martin, MD, PhD, Principal Investigator — Grupo G6
Locations (1):
- I.H. Hospital San Jose, Madrid, Madrid, Spain